CLINICAL TRIAL: NCT03057366
Title: A Phase 1 Study to Assess Mass Balance, Pharmacokinetics, and Metabolism of [14C]-Pevonedistat in Patients With Advanced Solid Tumors
Brief Title: A Study of [14 C]-Pevonedistat in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Pevonedistat-1013; U1111-1169-6648 (Registry Identifier: WHO); 2016-004132-37 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Results first posted 2019-05-08 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumors, Neoplasms, Advanced Solid
Keywords: Drug therapy
MeSH Terms: conditions — Neoplasms | interventions — pevonedistat; Docetaxel; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-Pevonedistat 25 mg/m^2 (Experimental): [14C]-pevonedistat (containing approximately 60-98 mCi [approximately 2.22-3.626 MBq] of radioactive tracer), infusion, intravenously, single dose on Day 1 of Week 1 in Part A. After completion of Part A, participants will have opportunity to continue into Part B. Participant will receive Pevonedistat 25 mg/m^2, infusion, intravenously, single dose on Days 1, 3 and 5 of each 21 day cycle, for up to 12 cycles along with docetaxel 75 mg/m^2, infusion, intravenously, over 1 hour on Day 1 of each 21 day cycle; or pevonedistat 20 mg/m^2, infusion, intravenously, single dose on Days 1, 3 and 5 of each 21 day cycle, for up to 12 cycles, followed by paclitaxel 175 mg/m^2, infusion, intravenously, over 3 hours along with carboplatin 20 mg/m^2, infusion, intravenously, over 30 minutes on Day 1 of 21 each cycle up to 12 cycles. Based on investigator and sponsor discretion, participants deriving benefits will continue to receive current combination therapy or pevonedistat alone beyond 12 cycles.
  Interventions: Drug: Pevonedistat; Drug: [14C]-Pevonedistat; Drug: Docetaxel; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Other Names: MLN4924; TAK-924
Drug: [14C]-Pevonedistat — [14C]-Pevonedistat intravenous infusion.
Drug: Docetaxel — Docetaxel intravenous infusion.
Drug: Carboplatin — Carboplatin intravenous infusion.
Drug: Paclitaxel — Paclitaxel intravenous infusion.

SUMMARY:
The purpose of this study is to assess the mass balance (that is, cumulative excretion of total radioactivity [TRA] in urine and feces) and to characterize the pharmacokinetics (PK) of pevonedistat in whole blood, plasma, and urine, and of TRA in plasma and whole blood following a single 1-hour infusion of 25 milligram per square meter (mg/m^2) [14C]-pevonedistat intravenous (IV) solution containing approximately 60 to 85 microcurie (mCi) (approximately 2.22-3.145 megabecquerel [MBq]) of TRA in participants with advanced solid tumors in Part A.

DETAILED DESCRIPTION:
The drug being tested in this study is called Pevonedistat. Pevonedistat is being tested to treat people with advanced solid tumors.

The study will enroll approximately 4 to 6 pharmacokinetics (PK)-evaluable participants in part A. After completion of the mass balance and absorption, distribution, metabolism, excretion (ADME) assessment in Part A of the study, eligible participants will have the opportunity to continue into Part B at a secondary study site, which would begin in approximately 2 weeks of completion of Part A.

* [14C]-Pevonedistat 25 mg/m^2
* Part B (optional): Pevonedistat in combination with chemotherapy regimens (Pevonedistat 25 mg/m^2 + docetaxel 75 mg/m^2 or pevonedistat 20 mg/m^2 + carboplatin 20 mg/m^2 + paclitaxel 175 mg/m^2)

All participants will receive study drug via intravenous route. This multi-center trial will be conducted in Hungary. Participants will remain confined to the study site for 9 to 14 days in Part A. Participation in Part B is optional, participants will be re-evaluated for inclusion/exclusion criteria before administrating treatment. Participants will undergo treatment in Part B for a maximum of 12 cycles (21 days cycle each) and will include approximately 36 weeks for Part A and B combined. Participants will attend an end of study visit 30 days after the last dose of study drug in both Part A and B.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed metastatic or locally advanced and incurable solid tumor that is felt to be appropriate for treatment with one of the 2 chemotherapy regimens in Part B of this study (carboplatin+paclitaxel or docetaxel), or have progressed despite prior standard therapy, or for whom conventional therapy is not considered effective. The tumor must be radiographically or clinically evaluable and/or measurable.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Expected survival longer than 3 months from enrollment in the study.
4. Recovered (that is, less than or equal to [<=] Grade 1 toxicity) from the effects of prior antineoplastic therapy.

Exclusion Criteria:

1. Has irregular defecation patterns (less than 1 defecation per 2 days or excessive diarrhea) and/or has a history of changes in bowel habits with daily routine or environment changes.
2. Prior treatment with radiation therapy involving greater than or equal to (>=) 25% of the hematopoietically active bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- Hungary (2):
  - Magyar Honvédség Egészségügyi Központ Onkológiai osztály, Budapest
  - PRA Magyarország Kft. Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Zhou X, Sedarati F, Faller DV, Zhao D, Faessel HM, Chowdhury S, Bolleddula J, Li Y, Venkatakrishnan K, Papai Z. Phase I study assessing the mass balance, pharmacokinetics, and excretion of [14C]-pevonedistat, a NEDD8-activating enzyme inhibitor in patients with advanced solid tumors. Invest New Drugs. 2021 Apr;39(2):488-498. doi: 10.1007/s10637-020-01017-x. Epub 2020 Oct 22. PMID 33089874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Hungary from 11 May 2017 to 05 November 2018.
Pre-assignment Details: Participants with advanced solid tumors were enrolled in this two-part study to receive intravenous infusion of pevonedistat in Part A and pevonedistat in combination with chemotherapy in Part B (optional part). One participant from Part A consented for Part B but did not meet the eligibility criteria and never received study treatment in Part B.
Groups:
- Part A: [14C]-Pevonedistat 25 mg/m^2: [14C]-pevonedistat (containing approximately 60-98 microcurie [mCi] [approximately 2.22-3.626 megabecquerel (MBq)] of radioactive tracer), infusion, intravenously, single dose on Day 1 of Week 1 in Part A.
- Part B: Pevonedistat + Paclitaxel and Carboplatin: Pevonedistat 20 mg/m^2, infusion, intravenously, single dose, on Days 1, 3 and 5 of each 21-days treatment cycle (up to 11 cycles), in combination with paclitaxel 175 mg/m^2, infusion, intravenously along with carboplatin AUC5, infusion, intravenously, on Day 1 of each 21-days treatment cycle (up to 11 cycles). Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
- Part B: Pevonedistat + Docetaxel: Pevonedistat 25 mg/m^2, infusion, intravenously, single dose on Days 1, 3 and 5 of each 21-days treatment cycle (up to 11 cycles), in combination with docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-days treatment cycle (up to 11 cycles). Pevonedistat was administered after the docetaxel chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Period: Part A
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2 | Part B: Pevonedistat + Paclitaxel and Carboplatin | Part B: Pevonedistat + Docetaxel
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2 | Part B: Pevonedistat + Paclitaxel and Carboplatin | Part B: Pevonedistat + Docetaxel
Started | 0 | 5 (Participants completed Part A, met eligibility criteria, and provided consent for Part B.) | 2 (Participants completed Part A, met eligibility criteria, and provided consent for Part B.)
Completed | 0 | 5 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A.
Groups:
- [14C]-Pevonedistat 25 mg/m^2: [14C]-pevonedistat (containing approximately 60-98 mCi [approximately 2.22-3.626 MBq] of radioactive tracer), infusion, intravenously, single dose on Day 1 of Week 1 in Part A. Participants who completed Part A and provided consent for Part B continued treatment in Part B. Participants received pevonedistat 20 mg/m^2, infusion, intravenously, single dose, on Days 1, 3 and 5 of each 21-days treatment cycle (up to 11 cycles), in combination with paclitaxel 175 mg/m^2, infusion, intravenously along with carboplatin AUC5, infusion, intravenously, on Day 1 of each 21-days treatment cycle (up to 11 cycles); or pevonedistat 25 mg/m^2, infusion, intravenously, single dose on Days 1, 3 and 5 of each 21-days treatment cycle (up to 11 cycles), in combination with docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 of each 21-days treatment cycle (up to 11 cycles). Pevonedistat was administered after the chemotherapies in Part B.
Arm/Group | [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The safety analysis set is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A.
  years | 61.8 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  Participants
    Female | 5
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 8
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 8
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  Participants
    Hungary | 8
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  kilogram (kg) | 82.38 (15.777)
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  centimeter (cm) | 165.9 (8.85)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  kilogram per square meter (kg/m^2) | 29.58 (4.674)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] — Population: The safety analysis set for Part A is defined as all enrolled participants who received at least 1 dose of [14 C]-pevonedistat during Part A. All safety analyses in Part A was performed using the safety population for Part A.
  square meter (m^2) | 1.943 (0.2195)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Cmax: Maximum Observed Plasma and Whole Blood Concentration for Pevonedistat
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The pharmacokinetic (PK) evaluable population included all enrolled participants who received the protocol-specified single [14C]-pevonedistat dose in Part A and did not receive any excluded medications throughout the completion of Part A and had sufficient concentration-time data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A: [14C]-Pevonedistat 25 mg/m^2: [14C]-pevonedistat (containing approximately 60-98 mCi [approximately 2.22-3.626 MBq] of radioactive tracer), infusion, intravenously, single dose on Day 1 of Week 1 in Part A.
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
nanogram per milliliter (ng/mL)
  Plasma | 234.3 (99.52)
  Whole blood | 6862.9 (1595.22)

2. Primary Outcome: Part A: Tmax: Time to Reach the Maximum Plasma and Whole Blood Concentration (Cmax) for Pevonedistat
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK evaluable population included all enrolled participants who received the protocol-specified single [14C]-pevonedistat dose in Part A and did not receive any excluded medications throughout the completion of Part A and had sufficient concentration-time data.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
hour
  Plasma | 0.980 [0.95 to 1.50]
  Whole Blood | 1.000 [0.98 to 1.53]

3. Primary Outcome: Part A: AUClast: Area Under the Plasma and Whole Blood Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Pevonedistat
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
hour*nanogram per milliliter (hr*ng/mL)
  Plasma | 1446.9 (374.46)
  Whole Blood | 59284.0 (10035.58)

4. Primary Outcome: Part A: Cmax: Maximum Observed Plasma and Whole Blood TRA Concentration for [14C]-Pevonedistat Drug-related Material
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram equivalent per milliliter
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
nanogram equivalent per milliliter
  Plasma | 293.6 (113.17)
  Whole Blood | 7336.6 (1270.99)

5. Primary Outcome: Part A: Tmax: Time to Reach the Maximum Plasma and Whole Blood TRA Concentration (Cmax) for [14C]-Pevonedistat Drug-related Material
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
hour
  Plasma | 0.980 [0.95 to 1.50]
  Whole Blood | 0.980 [0.98 to 2.00]

6. Primary Outcome: Part A: AUClast: Area Under the Plasma and Whole Blood TRA Concentration Curve From Time 0 to Time of the Last Quantifiable Concentration for [14C]-Pevonedistat Drug-related Material
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram equivalent per milliliter
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
hour*nanogram equivalent per milliliter
  Plasma | 3547.3 (1106.56)
  Whole Blood | 133259.0 (32678.72)

7. Primary Outcome: Part A: Aeurine,14C: Cumulative Amount of [14C]-Pevonedistat Excreted in Urine up to the Last Sampling Interval
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram equivalent (mcg eq)
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
microgram equivalent (mcg eq) | 19661.05 (4099.981)

8. Primary Outcome: Part A: Aefeces,14C: Cumulative Amount of [14C]-Pevonedistat Excreted in Feces up to the Last Sampling Interval
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg eq
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
mcg eq | 25029.45 (4333.04)

9. Primary Outcome: Part A: Aetotal,14C: Total Cumulative Excretion of [14C]-Pevonedistat From the Body
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg eq
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
mcg eq | 44690.50 (2090.833)

10. Primary Outcome: Part A: Aeurine: Cumulative Amount of Pevonedistat Dose Excreted in Urine at 144-168 Hours Post-dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
microgram (mcg) | 1161.47 (266.413)

11. Primary Outcome: Part A: Feurine: Cumulative Percentage of Pevonedistat Dose Excreted in Urine at 144-168 Hours Post-dose
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
percentage of dose | 2.45 (0.548)

12. Primary Outcome: Part A: Renal Clearance (CLR) for Pevonedistat
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
liter per hour (L/hr) | 0.8343 (0.27889)

13. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Part A: From first dose of study drug in Part A up to Day 31; Part B: From first dose of study drug in Part B up to Cycle 11 Day 35 (Cycle length is equal to [=] 21 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2 | Part B: Pevonedistat + Paclitaxel and Carboplatin | Part B: Pevonedistat + Docetaxel
Number analyzed (Participants) | 8 | 5 | 2
Participants
  TEAEs | 4 | 5 | 2
  SAEs | 1 | 2 | 1

14. Secondary Outcome: Part A: Percent Distribution of Total Radioactivity (TRA) for Pevonedistat and Its Metabolites in Plasma, Urine and Feces
Time Frame: Up to 168 hours post-dose
Population: The PK evaluable population included all enrolled participants who received the protocol-specified single [14C]-pevonedistat dose in Part A and did not received any excluded medications throughout the completion of Part A and had sufficient concentration-time data.
Measure: Mean (Standard Deviation); unit: percentage distribution of TRA
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2
Number analyzed (Participants) | 7
percentage distribution of TRA
  Pevonedistat in Plasma | 49.3 (9.8)
  Metabolite-1 in Plasma | 14.6 (4.9)
  Metabolite-2 in Plasma | 21.5 (3.0)
  Metabolite-3 in Plasma | 4.5 (0.6)
  Metabolite-7 in Plasma | 0.8 (0.3)
  Metabolite-10b in Plasma | 6.5 (2.1)
  Metabolite-16 in Plasma | 1.0 (0.4)
  Metabolite-22 in Plasma | 1.9 (0.8)
  Pevonedistat in Urine | 10.5 (6.1)
  Metabolite-1 in Urine | 46.5 (4.4)
  Metabolite-2 in Urine | 19.1 (2.1)
  Metabolite-3 in Urine | 9.9 (0.9)
  Metabolite-7 in Urine | 1.8 (0.7)
  Metabolite-10b in Urine | 3.5 (1.0)
  Metabolite-16 in Urine | 6.1 (2.5)
  Metabolite-22 in Urine | 1.3 (0.5)
  Metabolite-23 in Urine | 0.8 (0.2)
  Metabolite-24 in Urine | 1.7 (0.7)
  Pevonedistat in Feces | 30.3 (9.9)
  Metabolite-1 in Feces | 14.1 (8.3)
  Metabolite-2 in Feces | 34.0 (4.0)
  Metabolite-3 in Feces | 20.3 (2.9)
  Metabolite-7 in Feces | 1.3 (0.2)

15. Secondary Outcome: Part B: Number of Participants With Best Overall Response as Per Investigator's Assessment
Description: The best overall response was defined as the participants with best response among complete response (CR) or partial response (PR) or stable disease (SD), or progressive disease (PD). It was assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<) 10 millimeter (mm). PR: at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters as the best overall response after randomization. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to Cycle 11 (Cycle length =21 days)
Population: The response-evaluable population included all participants who received at least 1 dose of study drug in Part B, had measurable disease as entry criteria for Part B, and had at least 1 post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pevonedistat + Paclitaxel and Carboplatin | Part B: Pevonedistat + Docetaxel
Number analyzed (Participants) | 5 | 2
Participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 2 | 0
  PD | 3 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (From first dose of study drug in Part A up to Day 31; From first dose of study drug in Part B up to Cycle 11 Day 35)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Reported AEs and deaths are TEAEs that occurred between the first dose of the study drug and 30 days after the last dose of the study drug.
Arm/Group | Part A: [14C]-Pevonedistat 25 mg/m^2 | Part B: Pevonedistat + Paclitaxel and Carboplatin | Part B: Pevonedistat + Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/5 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/5 | 1/2
Other Adverse Events (participants affected / at risk) | 4/8 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: [14C]-Pevonedistat 25 mg/m^2 (N=8) | Part B: Pevonedistat + Paclitaxel and Carboplatin (N=5) | Part B: Pevonedistat + Docetaxel (N=2)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
FIBROSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: [14C]-Pevonedistat 25 mg/m^2 (N=8) | Part B: Pevonedistat + Paclitaxel and Carboplatin (N=5) | Part B: Pevonedistat + Docetaxel (N=2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (6) | 2 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (4)
Pain (General disorders) | 0 (0) | 2 (4) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (3)
Chest Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (7) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (6) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mueller's Mixed Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03057366/SAP_000.pdf
  • Study Protocol (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03057366/Prot_001.pdf